CLINICAL TRIAL: NCT00000799
Title: HPMPC (Cidofovir) Peripheral CMV Retinitis Trial Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Gilead Sciences (Industry)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: ACTG 281; GS-93-105; FDA 231A
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Cytomegalovirus Retinitis; HIV Infections
Keywords: Retinitis; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome; Antiviral Agents; cidofovir
MeSH Terms: conditions — Cytomegalovirus Retinitis; HIV Infections; Retinitis; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome | interventions — Cidofovir; Probenecid

INTERVENTIONS:
Drug: Cidofovir
Drug: Probenecid

SUMMARY:
To evaluate short-term and long-term safety and efficacy of intravenous cidofovir (HPMPC) for treatment of small peripheral cytomegalovirus (CMV) retinitis lesions. To provide data on the relative safety and efficacy of 2 doses of HPMPC as maintenance regimens.

DETAILED DESCRIPTION:
In Stage 1, up to 30 patients are randomized to either observation with deferral of treatment until the retinitis progresses (observation group), or to intravenous HPMPC at the higher dose for two consecutive weekly induction doses, followed by the lower dose every other week for maintenance. In Stage 2, up to 70 patients are randomized to observation or to HPMPC at the higher dose for two consecutive weekly induction doses followed by either dose every other week for maintenance, for a total of three treatment groups. Concomitant saline hydration and probenecid are administered to patients receiving HPMPC.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Oral trimethoprim/sulfamethoxazole.
* Aerosolized pentamidine.
* Dapsone.
* Fluconazole.
* Ketoconazole.
* Itraconazole.
* Rifabutin.
* Filgrastim (G-CSF).
* Antiretroviral agents.

Patients must have:

* AIDS by CDC criteria.
* CMV retinitis as determined by a SOCA-certified ophthalmologist, with lesion size, location, and severity as specified in the Disease Status field.

Prior Medication:

Allowed:

* Prophylaxis with anti-CMV agents.

Exclusion Criteria

Concurrent Medication:

Excluded:

* Ongoing therapy for CMV disease with ganciclovir, foscarnet, CMV hyperimmune immunoglobulin, or other investigational agents with anti-CMV activity.
* Therapy with nephrotoxic drugs, including amphotericin B, aminoglycoside antibiotics, vidarabine, and intravenous pentamidine.

Patients with the following prior conditions are excluded:

* History of renal disease or renal dialysis.
* History of clinically significant cardiac disease, including symptoms of ischemia, congestive heart failure, or arrhythmia.
* History of clinically significant probenecid allergy.

Prior Medication:

Excluded:

* Prior therapy for CMV disease with ganciclovir, foscarnet, CMV hyperimmune immunoglobulin, or other investigational agents with anti-CMV activity.
* Therapy with nephrotoxic drugs within the past 7 days, including amphotericin B, aminoglycoside antibiotics, vidarabine, and intravenous pentamidine.

Drug or alcohol abuse sufficient to hinder compliance with study.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Study Completion 1996-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - UCSD - Shiley Eye Ctr / SOCA, La Jolla, California
  - UCLA - Jules Stein Eye Institute / SOCA, Los Angeles, California
  - UCSF - San Francisco Gen Hosp, San Francisco, California
  - Northwestern Univ / SOCA, Chicago, Illinois
  - Johns Hopkins Hosp / SOCA, Baltimore, Maryland
  - New York Univ Med Ctr / SOCA, New York, New York
  - Univ of North Carolina / SOCA, Chapel Hill, North Carolina

REFERENCES:
- [Background] Parenteral cidofovir for cytomegalovirus retinitis in patients with AIDS: the HPMPC peripheral cytomegalovirus retinitis trial. A randomized, controlled trial. Studies of Ocular complications of AIDS Research Group in Collaboration with the AIDS Clinical Trials Group. Ann Intern Med. 1997 Feb 15;126(4):264-74. doi: 10.7326/0003-4819-126-4-199702150-00002. PMID 9036798